CLINICAL TRIAL: NCT04395157
Title: Optimizing Cognitive Remediation in VA Mental Health Rehabilitation Settings
Brief Title: Optimizing Cognitive Remediation
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: D3395-W; 1IK2RX003395 (NIH)
Record Dates: First submitted 2020-05-12; First posted 2020-05-20 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder; Mood Disorders
Keywords: Electroencephalography; Cognition; Rehabilitation
MeSH Terms: conditions — Schizophrenia; Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder; Mood Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Electrophysiological data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Veterans engaged in VA mental health rehabilitation/recovery: Veterans must be within 6 weeks of discharge from or current receive mental health treatment services in a VA San Diego Healthcare System psychosocial rehabilitation and recovery center (PRRC), mental health residential rehabilitation treatment program (RRTP), general mental health outpatient treatment, or recent acute mental health inpatient hospitalization.

SUMMARY:
Veterans with mental illness face challenges with community reintegration, including achieving vocational success, attaining their educational goals and going back to school, and maintaining a high quality of life. VA Mental Health Residential Rehabilitation Treatment Programs, Psychosocial Rehabilitation and Recovery Centers and other mental health treatment programs are designed to help Veterans overcome these barriers, but cognitive impairment often seen in Veterans with mental illness limits gains from these settings. Cognitive remediation interventions can be helpful, but they are either "one-size fits all," and thus may not be useful for all Veterans with mental illness, or are too narrow in scope, focusing on specific mental illnesses, limiting generalizability.

This project will test whether an objective neurophysiological biomarker, mismatch negativity (MMN), can better match the "right" Veteran to the "right" cognitive remediation treatment regardless of their specific mental health diagnosis.

DETAILED DESCRIPTION:
This is an observational, non-interventional study. Veterans with mental health diagnoses currently engaged in, or within 6 weeks of discharge from VA Mental Health Residential Rehabilitation Treatment Programs (RRTP), Psychosocial Rehabilitation and Recovery Centers (PRRC), and other mental health treatment settings (inpatient or outpatient mental healthcare) will be recruited. Veterans will have their cognitive functioning assessed. Following this, mismatch negativity (MMN) will be assessed via electroencephalography (EEG). Participants will undergo a 1 hour computerized cognitive training program. They will be interviewed about their attitudes about EEG and computerized cognitive training. They will be followed monthly for a total of 4 months from study entry to assess recovery trajectory. This study aims to enroll 104 Veterans from the VA San Diego Healthcare System.

The Specific Aims of this proposal are 1) Determine whether MMN is related to functioning, psychosocial recovery in VA rehabilitation milieus and programs; 2) Determine whether MMN is linked to cognition and predicts cognitive remediation exercise performance in a heterogeneous group of Veterans with mental illness. The proposal will also assess feasibility and acceptability of using biomarker-guided cognitive rehabilitation interventions in VA mental health rehabilitation settings.

Information gained from this study will help establish a precision-medicine approach towards cognitive rehabilitation for Veterans with mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Veterans are currently enrolled in or within 6 weeks of discharge from (as relevant): a VA San Diego Healthcare System (VASDHS) psychosocial rehabilitation and recovery center (PRRC), VASDHS mental health residential rehabilitation treatment program (RRTP), VASDHS acute inpatient hospitalization or VASDHS outpatient mental health treatment
* have a DSM-5 mental illness, including:

  * schizophrenia
  * schizoaffective disorder
  * delusional disorder
  * major depressive disorder
  * bipolar disorder
  * generalized anxiety disorder
  * PTSD
* fluent and literate in English
* no impairment in hearing or vision

Exclusion Criteria:

* active substance use within the last 30 days
* positive urine drug screen conducted as part of the screening process
* have acute/ongoing thoughts of self-harm or harming others
* intellectual disability or a neurocognitive disorder (i.e. dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans are currently enrolled in or within 6 weeks of discharge from (as relevant): a VA San Diego Healthcare System (VASDHS) psychosocial rehabilitation and recovery center (PRRC), VASDHS mental health residential rehabilitation treatment program (RRTP), VASDHS acute inpatient hospitalization or VASDHS outpatient mental health treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Mismatch Negativity (electrophysiological biomarker) | 3 months
  Mismatch negativity (micro-volts)
Cognition | 3 months
  Performance on MATRICS Consensus Cognitive Battery
Cognitive training performance | 3 months
  Performance on a 1 hour computerized cognitive training exercise
WHOQOL-BREF | 3 months
  Scores on the World Health Organization Quality of Life scale
WHODAS 2.0 | 3 months
  World Health Organization Disability Schedule 2.0

OTHER OUTCOMES:
Feasibility and acceptability of using biomarker-guided cognitive rehabilitation interventions in VA rehabilitation settings | 3 months
  Adapted Intrinsic Motivation Inventory (IMI) and Veteran qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Yash B. Joshi, MD PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT04395157/ICF_000.pdf